CLINICAL TRIAL: NCT06521541
Title: Whole Course Multi-model Prehabilitation to Improve Clinical Outcome in Patients Undergoing Neoadjuvant Treatment Prior to Gastrectomy : A Single Center Randomized Control Trial
Brief Title: Whole Course Multi-model Prehabilitation to Improve Clinical Outcome in Patients Undergoing Neoadjuvant Treatment Prior to Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prehab2024-01
Record Dates: First submitted 2024-07-14; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Prehabilitation
Keywords: Multimodal prehabilitation; Neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal prehabilitation group (Experimental): Patients received multimodal prehabilitation combined with ERAS before the gastrectomy.
  Interventions: Behavioral: Multimodal prehabilitation program
- ERAS group (Active Comparator): The ERAS pathway was followed in patients in the ERAS group.
  Interventions: Behavioral: ERAS program

INTERVENTIONS:
Behavioral: Multimodal prehabilitation program — Patients adopted planned, structural, repetitive and purposeful approach that includes elements of exercise, nutritional and psychological.Patients were evaluated for changes during neoadjuvant therapy and postoperative recovery
  Arms: Multimodal prehabilitation group
Behavioral: ERAS program — The core content is to adopt a series of optimized measures performed during the perioperative period on the basis of evidence-based medical findings to reduce the physiological and psychological stress of patients and to accelerate their recovery.
  Arms: ERAS group

SUMMARY:
The intention of research is to establish a multimodal prehabilitation protocol in patients who undergo neoadjuvant chemotherapy prior to gastrectomy, explore the feasibility and effectiveness of the measures and evaluate the effect of program on short-term clinical outcome, fitness and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2；
3. Endoscopic biopsies were pathologically confirmed as gastric adenocarcinoma；
4. The feasibility of neoadjuvant therapy was suggested by MDT, and the feasibility of radical gastrectomy was re-evaluated after neoadjuvant therapy;
5. Blood routine, liver function, kidney function, heart function and lung function were normal before neoadjuvant therapy, and there was no contraindication of chemotherapy and surgery;
6. The pregnancy test was negative within 1 month, and she was not pregnant or breastfeeding;
7. Informed consent and ability to comply with research protocols.

Exclusion Criteria:

1. metastasis;
2. End-stage cardiac insufficiency (LVEF<30% or NYHA class IV), liver cirrhosis (Child-Pugh classification C), End-stage renal failure (receives chronic dialysis), or ASA grade IV;
3. Cerebral hemorrhage, cerebral infarction, TIA or central nervous system disease or mental illness within 6 months, could not cooperate with the completion of neoadjuvant therapy and pre-rehabilitation exercise;
4. Patients have severe infections (such as MODS, etc.) or have allergic reactions to chemotherapy drugs and metabolic disorders;
5. Concurrent tumors or other diseases requiring simultaneous surgery (except laparoscopic gallbladder surgery);
6. Emergency surgery is required due to tumor complications (e.g., bleeding, perforation, obstruction);
7. Patients participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary capacity | Baseline (T0), Post-neoadjuvant chemotherapy (through completetion of neoadjuvant therapy, an average of 16 weeks), and prior to surgery(T2)
  The 6-minute walk test (6MWT) can be used to measure exercise capacity to reflect cardiopulmonary function.

SECONDARY OUTCOMES:
Patient's quality of life | Baseline (T0), Post-neoadjuvant chemotherapy (through completetion of neoadjuvant therapy, an average of 16 weeks), and prior to surgery(T2)
  QoL comprises patient-reported outcomes (PRO) of physical symptoms and psychosocial health status. Quality of Life Questionnaire (QLQ) C30 is sensitive tool for measuring individual performance status. Each index score ranges from 1 to 4, with higher scores indicating higher risk.
Serum albumin levels | Baseline (T0), Post-neoadjuvant chemotherapy (through completetion of neoadjuvant therapy, an average of 16 weeks), and prior to surgery(T2)
  The level of Serum albumin is used to assess nurtritional status.
sarcopenia | Baseline (T0), Post-neoadjuvant chemotherapy (through completetion of neoadjuvant therapy, an average of 16 weeks), and prior to surgery(T2)
  At the L3 level, total SM will be measured. Skeletal muscle index (SMI) will be calculated as follows: SM/height(m)2. SMI is used to assess nurtritional status.
completetion of neoadjuvant chemotherapy | Post-neoadjuvant chemotherapy (through completetion of neoadjuvant therapy, an average of 16 weeks)
  Discontinued due to adverse reactions
First exhaust and defecation | Postoperative (≤30 days after surgery)
  First exhaust and defecation is used to assess the postoperative recovery course.
First liquid diet | Postoperative (≤30 days after surgery)
  First liquid diet is used to assess the postoperative recovery course.
The incidence of postoperative complications | Postoperative (≤30 days after surgery)
  Refers to the incidence of early postoperative complications.
Duration of postoperative hospital stay | Postoperative (≤30 days after surgery)
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
Hospitalization costs | Postoperative (≤30 days after surgery)
  The expense from admission to discharge
3-year recurrence-free survival | 3 years
  3-year recurrence-free survival (RFS) rate
3-year overall survival | 3 years
  3-year overall survival (OS) rate

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Department of Gastrointestinal Surgery, Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR